CLINICAL TRIAL: NCT00227513
Title: A Phase I Study of Suberoylanilide Hydroxamic Acid (SAHA) in Combination With Bortezomib in Patients With Advanced Malignancies
Brief Title: Vorinostat and Bortezomib in Treating Patients With Metastatic or Unresectable Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00097; NCI-2009-00097 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000441195; H-2005-0205; CO 04906 (Other: University of Wisconsin Hospital and Clinics); 6910 (Other: CTEP); P30CA014520 (NIH); U01CA062491 (NIH)
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2013-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Bortezomib; Vorinostat

ARMS (1):
- Arm I (Experimental): Patients receive oral vorinostat (SAHA) twice daily on days 1-14 in step A. Patients receive oral vorinostat (SAHA) twice daily on days 1-4 and 8-11 in Step B and bortezomib IV over 3-5 seconds on days 2, 5, 9, and 12 during the first course and on days 1, 4, 8, and 11 during subsequent courses in both steps A and B. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Cohorts of 1-6 patients receive escalating doses of bortezomib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Up to 6 additional patients receive bortezomib at the MTD. Subsequent cohorts of 3-6 patients receive escalating doses of SAHA until the MTD of that drug is determined.
  Interventions: Drug: bortezomib; Drug: vorinostat

INTERVENTIONS:
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Drug: vorinostat — Given orally
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza

SUMMARY:
This phase I trial is studying the side effects and best dose of vorinostat and bortezomib in treating patients with metastatic or unresectable solid tumors. Drugs used in chemotherapy, such as vorinostat, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving vorinostat together with bortezomib may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of vorinostat (SAHA) and bortezomib in patients with metastatic or unresectable solid tumors.

SECONDARY OBJECTIVES:

I. Determine the pharmacokinetics and antitumor activity of this regimen in these patients.

II. Determine the toxic effects of this regimen in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive oral vorinostat (SAHA) twice daily on days 1-14 in step A. Patients receive oral vorinostat (SAHA) twice daily on days 1-4 and 8-11 in Step B and bortezomib IV over 3-5 seconds on days 2, 5, 9, and 12 during the first course and on days 1, 4, 8, and 11 during subsequent courses in both steps A and B. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 1-6 patients receive escalating doses of bortezomib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Up to 6 additional patients receive bortezomib at the MTD. Subsequent cohorts of 3-6 patients receive escalating doses of SAHA until the MTD of that drug is determined.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignancy, metastatic or unresectable disease
* Standard curative or palliative measures do not exist OR are no longer effective
* Measurable or evaluable disease
* No known brain metastases
* ECOG 0-2 OR Karnofsky 60-100%
* Life expectancy > 12 weeks
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* No history of myocardial infarction
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No severe pulmonary disease requiring oxygen
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 28 days after study participation
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to study drugs or agents
* No pre-existing neuropathy ≥ grade 2
* No uncontrolled illness
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No prior radiotherapy to > 25% of bone marrow
* At least 4 weeks since prior radiotherapy and recovered
* At least 2 weeks since prior valproic acid
* No prior bortezomib
* No concurrent enzyme-inducing anticonvulsant agents
* No other concurrent investigational agents
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2005-07; Primary Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) determined according to dose-limiting toxicities (DLTs) graded using Common Terminology Criteria for Adverse Events version 3.0 (CTCAE v3.0) | 21 days
Frequency and severity of toxicity incidents assessed by Common Terminology Criteria for Adverse Events version 3.0 (CTCAE v3.0) | Up to 5 years

SECONDARY OUTCOMES:
Anti-tumor activity by tumor measurements assessed by RECIST | Up to 5 years
Peak plasma concentration (Cmax) of SAHA | Days 1, 2, and 12
Time to SAHA Cmax (Tmax) | Days 1, 2, and 12
Clearance of SAHA | Days 1, 2, and 12

CONTACTS AND LOCATIONS:
Overall Officials: George Wilding, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States